CLINICAL TRIAL: NCT04260737
Title: Developing and Testing an Interactive Decision Aid for Newly Diagnosed Prostate Cancer Patients
Brief Title: Interactive Decision Aid for Men Diagnosed With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reykjavik University (Other)
Collaborators: The Icelandic Research Fund (Unknown); The Icelandic Cancer Society (Unknown)
Responsible Party: Principal Investigator, Dr. Heiddis B Valdimarsdottir, Professor, Reykjavik University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VSN-18-127; 141490-052 (Other Grant/Funding Number: The Icelandic Research Fund)
Record Dates: First submitted 2020-01-08; First posted 2020-02-07 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Prostate Cancer
Keywords: Localized Prostate Cancer; Decision Aid; Medical Decision Making
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Decision Support Techniques; Menogaril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): The control group will receive standard care for localized prostate cancer, i.e., information from their doctor and an information brochure.
- Decision Aid + Standard Care (Experimental): The intervention group will receive standard care and intervention that includes a website with the Decision Aid which covers the following:
  1. An overview about prostate cancer;
  2. An overview of different treatment options (e.g. surgery and active surveillance)
  3. The pros and cons of different treatment options (e.g., physical, emotional, social).
  4. A value clarification exercise that is designed to assist participants to weigh the pros and cons of each prostate cancer management option.
  Interventions: Other: Decision Aid for Men with Localized Prostate Cancer

INTERVENTIONS:
Other: Decision Aid for Men with Localized Prostate Cancer — The intervention is an interactive decision aid aimed to assist newly diagnosed prostate cancer patients with their treatment management options.
  Arms: Decision Aid + Standard Care

SUMMARY:
Prostate cancer is the second leading cause of cancer related deaths in the western world (National Cancer Institute, 2011). Prostate cancer diagnosis relates to significant psychological distress (Roesch et al, 2005; Hervouet et al, 2005). The management options available for men with localized prostate cancer typically offer similar survival rate and one treatment has not been determined more effective than other. Variance in severity, duration and frequency of side effects between treatments is considerable (National Cancer Institute, 2011). This can make the choice between management options challenging and distressing. Researches show that patients that are actively involved and provided with sufficient information have better health outcomes (Stewart, 1995).

The study involves implementing interactive, web-based decision-aid to assist men with localized prostate cancer with their decision regarding their prostate cancer management options. Participants will be randomized to standard-care (SC) and SC + interactive decision-aid (IDA). The SC group will meet with their urologist and receive and information brochure. In addition the IDA group will receive a website that includes a wealth of information (e.g., overview about prostate cancer, overview of different treatment options, pros and cons of different treatment options and a value clarification exercise that is designed to assist participants to weigh the risks and benefits of each prostate cancer management option).

The effectiveness of the intervention will be evaluated with questionnaires administered prior to randomization (baseline) and then again two weeks, one, three and six months after the randomization.

Aim 1. Evaluate the relative impact of SC versus SC + IDA on medical decision making. It is hypothesized that participants randomized to the SC + IDA arms will have improved decision making (e.g., reduced decisional conflict) and psychosocial outcomes (e.g., distress), compared to those randomized to SC only.

Aim 2. Identify mechanisms by which the interventions impact patient outcomes. It is hypothesized that: 1) improved decision making and psychosocial outcomes for the IDA arms will be mediated by increased knowledge; 2) participants who are undecided about the treatment decision and those that have information-seeking decision styles will benefit most from the decision-aid interventions.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with localized prostate cancer.

Exclusion Criteria:

* Reads and understands Icelandic
* Can give informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only those that have been assigned the biological sex of male at birth are eligible.
Enrollment: 163 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change in decisional conflict over time | Baseline, 2 weeks, 1 month, 3 months and 6 months.
  The Decisional Conflict Scale (DCS) is a measure that was designed to evaluate health-care-consumer decisions. It is a 16-item measure and the answers range from "strongly agree" to "strongly disagree" on a five point Likert scale. Scores on DCS range from 0 to 100, were higher score indicate greater decisional conflict. It has test-retest reliability of 0.81 and internal consistency ranges from α=.0.78 to 0.92.
Change in decisional regret over time | 2 weeks, 1 month, 3 months and 6 months.
  The Decision Regret Scale (DRS) measures regret after health care decision. It is a 5-item measure and the answers range from "strongly agree" to "strongly disagree" on a five point Likert scale. Scores on DRS range from 0 to 100, were higher score indicate more regret after health care decision. It has good internal consistency that ranges from α=.0.81 to 0.92.
Change in satisfaction with decision over time | 2 weeks, 1 month, 3 months and 6 months.
  The Satisfaction with Decision Scale (SWDS) measures satisfaction with health care decision. It is a 5-item measure and the answers range from "strongly agree" to "strongly disagree" on a five point Likert scale. Scores on SWDS range from 5 to 25, were higher score indicate more satisfaction with a decision.The scale has good internal consistency (α=.0.86).
Change in anxiety over time | Baseline, 2 weeks, 1 month, 3 months and 6 months.
  The Generalized Anxiety Disorder - 7 (GAD-7) is a 7-item measure used to screen for general anxiety disorder and to measure its severity. It is also a good screening tool for social anxiety disorder, panic disorder and post traumatic stress disorder. Response options range from "not at all" to "several days" on a 4-point Likert scale. GAD-7 total score ranges from 0 to 21, were higher score indicates more severe anxiety. It has excellent internal consistency (α = 0.92).
Change in depression over time | Baseline, 2 weeks, 1 month, 3 months and 6 months.
  The Patient Health Questionnaire (PHQ-9) is a widely used and well validated measure used to screen for depression and assess severity of it. It is a 9-item scale and answers are on 4-point Likert scale ranging from "not at all" to "nearly every day". PHQ-9 total score ranges from 0 to 27, were higher score indicates more severe depression. PHQ-9 has been shown to be a reliable and valid measure.
Change in Stress over time | Baseline, 2 weeks, 1 month, 3 months and 6 months.
  The Perceived Stress Scale (PSS-10) is a 10-item scale used to measure stress. Each item on the list is rated on a five point Likert scale ranging from "never" to "very often". PSS-10 total score ranges from 0 to 40, were higher score indicates higher perceived stress. The PSS has adequate reliability and validity.
Change in Stress over time | Baseline, 2 weeks, 1 month, 3 months and 6 months.
  The NCCN Distress Thermometer and checklist is a widely used screening measure for distress in cancer patients. It consists of a distress thermometer where participants assess their distress on a scale from 0 to 10, were 0 indicates no distress and 10 extreme distress. Additionally participants answer a problem checklist with several domains to identify what area of life distresses the participant.
Change in Cancer related Stress over time | Baseline, 2 weeks, 1 month, 3 months and 6 months.
  The Impact of events scale-revised (IES-R) is a widely used questionnaire that measures trauma related stress, that is cancer specific distress. It is a 22-item measure that includes three factors; avoidance, hyper arousal and intrusion. Those factors together form a cancer-specific distress measure and the higher the score on the scale suggest more distress. Total score range from 0 to 88. The IES-R has high internal consistency and test-retest reliability ranges from 0.51-0.94.

SECONDARY OUTCOMES:
Control preference | Baseline
  The control preference scale (CPS) assesses the patient's preferred role in the decision-making process. It measures how people with life-threatening illnesses make treatment decisions. It measures the degree of control a person wants to have when making a medical treatment management decision.The scale is a single item and displays five possible roles of patient in decision making, that is fully passive, semi-passive, collaborative, semi-active and fully active.
Localized Prostate cancer knowledge | Baseline, 2 weeks, 1 month, 3 months and 6 months.
  The localized prostate cancer knowledge scale is a 9-item list that assesses participants knowledge of localized prostate cancer and prostate cancer management options. The scale was developed for this study based on method used by Berger, Grønberg, Loge, Kaasa and Sand (2018). Total score range from 0 to 9, were higher score indicates better knowledge of localized prostate cancer and prostate cancer management options.
Health Information Orientation | Baseline
  The Health Information Orientation Scale (HIOS) measures underlying reasons for avoiding or seeking information in health context. The scale consists of 8 items and has two factors, that is information engagement and information apprehension. Both factors show adequate construct validity and reliability. Total score range from 0 to 32, were higher score indicates greater information apprehension and information engagement.
Intolerance of uncertainty | Baseline
  The Intolerance of uncertainty-12 (IUS-12) measures response to ambiguous situation and uncertainty. The scale consists of 12 items. Total score range from 12 to 60, where higher score indicates greater intolerance of uncertainty. The IUS shows good psychometric properties.

CONTACTS AND LOCATIONS:
Overall Officials: Heiddis B Valdimarsdottir, PhD, Principal Investigator — Reykjavik University; Birna Baldursdottir, PhD, Study Director — Reykjavik University
Locations (1):
- Reykjavik University, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roesch SC, Adams L, Hines A, Palmores A, Vyas P, Tran C, Pekin S, Vaughn AA. Coping with prostate cancer: a meta-analytic review. J Behav Med. 2005 Jun;28(3):281-93. doi: 10.1007/s10865-005-4664-z. PMID 16015462
- [Background] Hervouet S, Savard J, Simard S, Ivers H, Laverdiere J, Vigneault E, Fradet Y, Lacombe L. Psychological functioning associated with prostate cancer: cross-sectional comparison of patients treated with radiotherapy, brachytherapy, or surgery. J Pain Symptom Manage. 2005 Nov;30(5):474-84. doi: 10.1016/j.jpainsymman.2005.05.011. PMID 16310621
- [Background] Stewart MA. Effective physician-patient communication and health outcomes: a review. CMAJ. 1995 May 1;152(9):1423-33. PMID 7728691
- [Background] Berger O, Gronberg BH, Loge JH, Kaasa S, Sand K. Cancer patients' knowledge about their disease and treatment before, during and after treatment: a prospective, longitudinal study. BMC Cancer. 2018 Apr 3;18(1):381. doi: 10.1186/s12885-018-4164-5. PMID 29614997